CLINICAL TRIAL: NCT00729053
Title: A Phase 2, Multi-Center, Randomized, Open-Label Study of Two Dose Levels of IMOxine® (IMO-2055 for Injection) in Patients With Metastatic or Locally Recurrent Clear Cell Renal Carcinoma
Brief Title: Study of IMO-2055 in Metastatic or Locally Recurrent Clear Cell Renal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2055-003
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Renal Cell Carcinoma
Keywords: renal; cell; renal carcinoma; metastatic; recurrent; treatment naive
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Recurrence | interventions — IMO-2055

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Previous treatment, 0.16mg/kg (Active Comparator): Patients will have clear cell renal carcinoma with previous treatment. Patients will receive weekly SC injections of IMO-2055 at a dose of 0.16mg/kg
  Interventions: Drug: IMO-2055
- Previous treatment, 0.64mg/kg (Active Comparator): Patients will have clear cell renal carcinoma with previous treatment. Patients will receive weekly SC injections of IMO-2055 at a dose of 0.64mg/kg
  Interventions: Drug: IMO-2055
- Treatment Naive, 0.16mg/kg (Active Comparator): Patients will have clear cell renal carcinoma without previous treatment. Patients will receive weekly SC injections of IMO-2055 at a dose of 0.16mg/kg
  Interventions: Drug: IMO-2055
- Treatment Naive, 0.64mg/kg (Active Comparator): Patients will have clear cell renal carcinoma without previous treatment. Patients will receive weekly SC injections of IMO-2055 at a dose of 0.64mg/kg
  Interventions: Drug: IMO-2055

INTERVENTIONS:
Drug: IMO-2055 — immunostimulatory oligonucleotide

SUMMARY:
* Multi-Center
* Randomized
* Open-Label Study of single agent IMO-2055
* Patients who have Metastatic or Locally Recurrent Clear Cell Renal Carcinoma (RCC)

DETAILED DESCRIPTION:
This is a study of 2 dose levels (0.16 or 0.64 mg/kg) of IMO-2055 administered by weekly subcutaneous (SC) injections in two patient populations, treatment naïve or previously treated patients. Each dose group (treatment naive or previously treated) will be randomized to receive one of the 2 doses being studied.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV clear cell renal carcinoma with metastatic or locally recurrent disease that is not surgically resectable.
* At least one measurable lesion
* Adequate organ function
* Any prior treatment of renal cell cancer was concluded at least 4 weeks prior.
* If female and of childbearing potential, a negative serum pregnancy test performed and documented no more than 14 days before the first dose of study drug.

Exclusion Criteria:

* Known untreated central nervous system (CNS) metastasis
* Pre-existing autoimmune or antibody-mediated diseases
* Other significant medical disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-06; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bexon, MD, Study Director — Idera Pharmaceuticals
Locations (1):
- Georgetown University, Lombardi Cancer Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
Started | 23 | 23 | 23 | 23
Completed | 23 | 23 | 23 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg | Total
Number analyzed (Participants) | 23 | 21 | 22 | 23 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years at the time of screening.
  Years | 60.1 (10.6) | 59.2 (10.3) | 65.6 (9.4) | 60.6 (12.0) | 61.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 11 | 8 | 31
  Male | 13 | 19 | 11 | 15 | 58

OUTCOME MEASURES:

1. Primary Outcome: Best Response by RECIST v1.0
Description: Best overall objective (i.e., radiological) response by RECIST v1.0 for target lesions: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR in patients with clear cell metastatic or locally recurrent renal cell carcinoma treated with IMO-2055.
Time Frame: From start of treatment every 8 weeks (every 2 cycles), 1 month post-treatment, then every 3 months (up to 1 year) until documented disease progression or initiation of an alternative therapeutic treatment regimen.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
Number analyzed (Participants) | 23 | 21 | 22 | 23
Participants | 0 | 1 | 0 | 1

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) by National Cancer Institute (NCI) Grade/Severity
Description: Number of patients with Treatment-emergent adverse events (TEAEs) by National Cancer Institute (NCI) grade/severity that began on or after the date of the first injection of study drug or worsened in severity or frequency after study drug was administered.
Time Frame: From start of treatment through one month after the end of study visit (up to 28 weeks)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
Number analyzed (Participants) | 23 | 23 | 23 | 23
Participants
  Patients with at least 1 TEAE | 23 | 23 | 21 | 22
  Patients with at least 1 serious TEAE | 6 | 10 | 5 | 8
  Patients with a TEAE related to treatment | 21 | 22 | 16 | 19
  Patients with at least 1 severe (Grade+) TEAE | 9 | 14 | 6 | 11

3. Secondary Outcome: Duration of Response by RECIST v1.0
Description: Time in days from the date of the first response by RECIST v1.0 to documented disease progression or death from any cause.
Time Frame: Every 8 weeks (2 cycles) from first response to documented disease progression during treatment, 1 month post-treatment, then every 3 months (up to 1 year) until documented disease progression or initiation of an alternative therapeutic treatment regimen.
Population: Participants with reported response as reflected in Outcome Measure 1
Measure: Number; unit: Days
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
Number analyzed (Participants) | 0 | 1 | 0 | 1
Days |  | 179 |  | 52

4. Secondary Outcome: Overall Survival at 1 Year
Description: Overall survival is defined as (date of death +1 - date of randomization). Patients without an event (death) during treatment or follow-up will have their date censored on the last visit the patient was known to be alive.
Time Frame: From date of randomization until the date of progression or date of death from any cause, whichever came first, asses up to 1 year after the last dose of study drug.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
Number analyzed (Participants) | 23 | 21 | 22 | 23
Participants | 15 | 14 | 14 | 15

5. Secondary Outcome: Time to Disease Progression.
Description: Time between the date of randomization to the Study Day of documented disease progression (an increase in tumor burden of at least 20%, appearance of new lesions, or unequivocal progression of non-measurable disease) or death (whichever comes first) by RECIST v1.0. Patients who had not progressed at last disease assessment, but whose progression status was unknown at the date last known alive, date of death, or date of study exit (whichever comes first), had event time censored at the date of last assessment. Patients who did not die and did not progress during treatment or follow-up had their event time censored on the last contact date.
Time Frame: Every 8 weeks (2 cycles) during the study and every 3 months for 1 year until documented disease progression
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
Number analyzed (Participants) | 23 | 21 | 22 | 23
Days | 103.0 [56.0 to 123.0] | 131.0 [60.0 to 178.0] | 138.5 [108.0 to 217.0] | 59.0 [53.0 to 123.0]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 30 days after the final dose of study drug (up to 28 weeks).
Description: Treatment-Emergent AEs were defined as those events which were not present at the pre-study evaluation, or worsened in severity after the start of treatment. Any AEs starting after study completion or withdrawal were not tabulated.
Arm/Group | Previous Treatment, 0.16mg/kg | Previous Treatment, 0.64mg/kg | Treatment Naive, 0.16mg/kg | Treatment Naive, 0.64mg/kg
All-Cause Mortality (participants affected / at risk) | 0/23 | 1/23 | 1/23 | 1/23
Serious Adverse Events (participants affected / at risk) | 6/23 | 10/23 | 5/23 | 8/23
Other Adverse Events (participants affected / at risk) | 23/23 | 23/23 | 21/23 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Treatment, 0.16mg/kg (N=23) | Previous Treatment, 0.64mg/kg (N=23) | Treatment Naive, 0.16mg/kg (N=23) | Treatment Naive, 0.64mg/kg (N=23)
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 4 | 1 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Adverse drug reaction (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 2
Chest pains (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Hypertenisve heart disease (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdomen wall abcess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure, acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Anticoagulant above therapeutic range (Investigations) | 0 | 0 | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Mental status change (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Treatment, 0.16mg/kg (N=23) | Previous Treatment, 0.64mg/kg (N=23) | Treatment Naive, 0.16mg/kg (N=23) | Treatment Naive, 0.64mg/kg (N=23)
Fatigue (General disorders) | 14 | 13 | 11 | 9
Nausea (Gastrointestinal disorders) | 14 | 12 | 6 | 10
Chills (General disorders) | 8 | 16 | 7 | 10
Headache (Nervous system disorders) | 10 | 7 | 9 | 8
Pyrexia (General disorders) | 3 | 13 | 5 | 9
Vomiting (Gastrointestinal disorders) | 7 | 7 | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 5 | 5
Constipation (Gastrointestinal disorders) | 4 | 6 | 1 | 8
Diarrhea (Gastrointestinal disorders) | 4 | 7 | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 5 | 6 | 2 | 4
Anemia (Blood and lymphatic system disorders) | 4 | 3 | 5 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 2 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 5 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 3
Peripheral edema (General disorders) | 2 | 3 | 1 | 4
Insomnia (Psychiatric disorders) | 3 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other